CLINICAL TRIAL: NCT01543789
Title: The Flemish Umbilical Nitinol Mesh Trial, a Multicenter Randomized Controlled Trial.
Brief Title: The Flemish Umbilical Nitinol Mesh Trial, a Multicenter Trial
Acronym: FUN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Medri (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC/2012/072
Record Dates: First submitted 2012-02-10; First posted 2012-03-05 (Estimated); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Umbilical Hernia
Keywords: Umbilical Hernia
MeSH Terms: conditions — Hernia, Umbilical

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intraperitoneal mesh placement (Experimental): Mesh placement inside the peritoneal cavity
  Interventions: Procedure: Intraperitoneal mesh placement
- Preperitoneal mesh placement (Active Comparator): Mesh placement between peritoneum and muscle layer.
  Interventions: Procedure: Preperitoneal mesh placement

INTERVENTIONS:
Procedure: Intraperitoneal mesh placement — Mesh placement inside the peritoneal cavity.
  Arms: Intraperitoneal mesh placement
Procedure: Preperitoneal mesh placement — Mesh placement between peritoneum and muscle layer.
  Arms: Preperitoneal mesh placement

SUMMARY:
The use of mesh in the repair of umbilical hernias is a gold standard. The best location of the mesh remains a matter of discussion, i.e. it might be placed inside the peritoneal cavity (open intraperitoneal onlay mesh) or between the peritoneum and the muscle layers, so not in contact with the viscera (retromuscular or preperitoneal). The Rebound mesh consists of polypropylene, i.e. the most used fabric for meshes, in combination with a nitinol memory ring. This ring allows the surgeon to position the mesh more flat, with less wrinkling and subsequently better tissue ingrowth. It also saves time for both patient's anesthesia and the surgery.

This type of mesh (one coated with PTFE for intra-abdominal use and one pure polypropylene for preperitoneal use), will be used in this multicentric trial, to evaluate the best procedure in terms of efficacy, safety and postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent from the patient or his/her legal representative
* primary umbilical hernia requiring elective surgical repair
* diameter between 0 and 3 cm

Exclusion Criteria:

* no written informed consent
* incisional hernia at the level of the umbilicus
* recurrent umbilical hernia, as they have to be considered an incisional hernia
* emergency surgery (incarcerated hernia)
* pregnancy
* non-compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-03; Primary Completion 2015-12 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Operation time between preperitoneal mesh placement versus intraperitoneal mesh placement. | Total duration of the operation with an expected average of approximately 45 minutes.
  Time registration of the operating time will be extracted from the hospital electronic patient files.

SECONDARY OUTCOMES:
Surgical wound morbidity complication rate. | Up to 1 year.
Recurrence Rate | up to 2 years
  Clinical examination will be performed. No ultrasound, unless doubt about recurrence.
Pain evaluation | within 2 weeks prior to surgery, after 4 weeks, after 1 year and after 2 years
  A questionnaire and Visual Analog Scale (VAS) will be filled out. The patient is asked whether he or she has pain. Answer NO: VAS = 0, Yes: patient will determine the exact VAS score.
Discomfort evaluation. | Within 2 weeks prior to surgery, after 4 weeks, after 1 year and after 2 years.
  A questionnaire and Visual Analog Scale (VAS) will be filled out. The patient is asked whether he or she has discomfort. Answer NO: VAS = 0, Yes: patient will determine the exact VAS score.

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Berrevoet, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (3):
- Belgium (3):
  - ASZ Aalst, Aalst
  - Ghent University Hospital, Ghent
  - UZ Leuven, Leuven

REFERENCES:
- See also: Related Info — http://www.uzgent.be